CLINICAL TRIAL: NCT00054886
Title: Phase II Study Of Single-Agent SU011248 In The Second-Line Treatment Of Patients With Metastatic Renal Cell Carcinoma
Brief Title: Study of the Safety and Efficacy of SU-011,248 in Adult Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTKC-0511-014
Record Dates: First submitted 2003-02-12; First posted 2003-02-13 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2006-07

CONDITIONS: Kidney Neoplasms
MeSH Terms: conditions — Kidney Neoplasms

INTERVENTIONS:
Drug: SU-011,248

SUMMARY:
The primary goal of the study is to evaluate the effectiveness and safety of SU-011,248 as a treatment for metastatic kidney cancer.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must be at least 18 years of age with a diagnosis of metastatic kidney cancer.
* The patient's kidney cancer must have gotten worse during/after previous cytokine-based therapy was given.
* Any side effects from prior therapy must have subsided, and blood and urine tests must show adequate bone marrow, liver, and kidney function

Exclusion Criteria:

* Prior treatment with any systemic therapy other than 1 prior cytokine-based treatment regimen;
* Prior surgical resection of or irradiation to the only site of measurable disease;
* Ongoing severe hematuria;
* Other active second malignancy;
* Cardiovascular diseases or conditions within the last 12 months;
* Known brain metastases;
* Known HIV-positive or AIDS-related illness;
* Pregnant or breast-feeding women;
* Current participation in other clinical trials;
* Other severe acute or chronic medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63
Dates: Start 2003-01; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was overall response rate (ORR) and the ORR achieved for the study was 40%.

SECONDARY OUTCOMES:
The secondary endpoints included time to progression (TTP) and overall survival (OS). The median TTP for the study was 8.7 months and the median OS was 16.4 months. SU011248 was generally well tolerated.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Mission Hills, California
  - Pfizer Investigational Site, Monterey Park, California
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Madison, Wisconsin

REFERENCES:
- [Derived] de Velasco G, McKay RR, Lin X, Moreira RB, Simantov R, Choueiri TK. Comprehensive Analysis of Survival Outcomes in Non-Clear Cell Renal Cell Carcinoma Patients Treated in Clinical Trials. Clin Genitourin Cancer. 2017 Dec;15(6):652-660.e1. doi: 10.1016/j.clgc.2017.03.004. Epub 2017 Mar 21. PMID 28410911
- [Derived] Grunwald V, Lin X, Kalanovic D, Simantov R. Early Tumour Shrinkage: A Tool for the Detection of Early Clinical Activity in Metastatic Renal Cell Carcinoma. Eur Urol. 2016 Dec;70(6):1006-1015. doi: 10.1016/j.eururo.2016.05.010. Epub 2016 May 26. PMID 27238653
- [Derived] Grunwald V, McKay RR, Krajewski KM, Kalanovic D, Lin X, Perkins JJ, Simantov R, Choueiri TK. Depth of remission is a prognostic factor for survival in patients with metastatic renal cell carcinoma. Eur Urol. 2015 May;67(5):952-8. doi: 10.1016/j.eururo.2014.12.036. Epub 2015 Jan 7. PMID 25577718
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=RTKC-0511-014&StudyName=Study+of+the+Safety+and+Efficacy+of+SU%2D011%2C248+in+Adult+Patients+With+Advanced+Kidney+Cancer